CLINICAL TRIAL: NCT03273036
Title: Comparison of Perioperative Outcome Between Corticosteroids and Placebo in Transforaminal Endoscopic Lumbar Discectomy. A Single-center Randomized Placebo-controlled Trial.
Brief Title: Perioperative Outcome of Corticosteroids in Transforaminal Endoscopic Lumbar Discectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Jatupon Kongtharvonskul, principle investigator, Ramathibodi Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ID 03-54-23
Record Dates: First submitted 2017-08-29; First posted 2017-09-06 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- epidural steroid injection (Active Comparator): 40 mg triamcinolone acetate 1 cc
  Interventions: Drug: 40 mg Triamcinolone acetate 1 cc
- placebo injection (Placebo Comparator): no injection agent
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: 40 mg Triamcinolone acetate 1 cc — 40 mg Triamcinolone acetate 1 cc
  Arms: epidural steroid injection
Drug: Placebos — no injected agent
  Arms: placebo injection

SUMMARY:
The endoscopic discectomy has rapidly developed and increased need by patients. This procedure is widely performed by interventional pain physicians as well as by spine surgeons because it requires no general anesthesia or admission to a hospital. Many studies were reported that corticosteroid injection can inhibit persistent postoperative pain in lumbar discectomy. However, data of perioperative epidural steroids after an endoscopic discectomy is lacking.

DETAILED DESCRIPTION:
To examine whether corticosteroid administered epidural space in patients undergoing endoscopic lumbar discectomy reduces postoperative morphine consumption, back and leg pain relief, improves functional disability comparing to placebo

ELIGIBILITY:
Inclusion Criteria:

* Lumbar disc herniation patient age 20-45 year-old who have symptom duration was at least 6 weeks and conservative treatment failed

Exclusion Criteria:

* Refuse to participate and inform consent, Previous spinal surgery, History of allergic to steroid

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2015-05-01 (Actual); Study Completion 2015-05-01 (Actual)

PRIMARY OUTCOMES:
Post-operative morphine consumption | Post operative 24 hour of morphine consumption in mg

SECONDARY OUTCOMES:
Visual analog score (back and leg) 0-10 | 1 day, 2, 6 ,12, 24 weeks
Oswestry disability index (ODI | 2, 6 ,12, 24 weeks
MacNab scores | 2, 6 ,12, 24 weeks

IPD SHARING:
Plan to Share IPD: No